CLINICAL TRIAL: NCT05546827
Title: PRISAM: Pre-Operative Radiotherapy and Immunotherapy for Sinonasal and Anorectal Melanoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0330; NCI-2022-07760 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2022-09-15; First posted 2022-09-21 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Sinonasal Melanoma; Anorectal Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sinonasal melanoma: patients with sinonasal melanoma (Experimental): A. Patients with upfront resectable disease
  Treatment:
  * Immunotherapy
  * 20 fraction radiation therapy +/- ongoing immunotherapy
  * Surgery
  B. Patients whose disease is not resectable at presentation
  Treatment:
  Immunotherapy with potential to enter resectable disease pathway if tumor becomes resectable or continue treatment as per multidisciplinary team preference if tumor does not become resectable
  Interventions: Procedure: Surgical resection
- Anorectal melanoma: patients with anorectal melanoma (Experimental): A. Patients with disease resectable with a sphincter sparing procedure
  Treatment:
  * Immunotherapy
  * 5 fraction radiation therapy
  * Surgery
  B. Patients with disease not resectable with a sphincter sparing procedure
  Treatment:
  * Immunotherapy to maximal response
  * 5 or 15 fraction radiation (depending on immunotherapy response) +/- ongoing immunotherapy
  * Surgery or biopsy
  Interventions: Procedure: Surgical resection

INTERVENTIONS:
Procedure: Surgical resection — Surgical resection after receiving neodjuvant combination immunotherapy followed by radiation therapy.

SUMMARY:
The goal of this clinical research study is to learn if pre-operative radiation therapy after starting immune checkpoint inhibition can help patients with sinonasal or anorectal melanoma have better outcomes

DETAILED DESCRIPTION:
To determine the rate of pathologic response (<50% viable tumor or >50% fibrosis) for non-metastatic sinonasal melanoma patients having surgical resection after receiving neoadjuvant combination immunotherapy followed by radiation therapy.

To determine the rate of pathologic response (<50% viable tumor or >50% fibrosis) for non-metastatic anorectal melanoma patients receiving neoadjuvant intent combination immunotherapy followed by radiation therapy.

ELIGIBILITY:
Inclusion Criteria

For all patients

* Evidence of mucosal tumor on clinical exam or imaging.
* No evidence of distant metastasis
* Patients must be planned for combination immunotherapy (e.g. ipilimumab and nivolumab or nivolumab and relatlimab).
* ECOG performance status ≤3.
* Age ≥18 years because melanoma is extremely rare in patients <18 years of age and RT is considered high risk in this population due to risk of secondary malignancy and potentially growing tissues that may be adversely impacted by RT.
* RT is a known teratogen. For this reason women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. (refer to MDA Policy CLN 1114) This includes all female patients, between the onset of menses and 55 years unless the patient presents with an applicable exclusionary factor which may be one of the following:
* Postmenopausal (no menses in greater than or equal to 12 consecutive months).
* History of hysterectomy or bilateral salpingo-oophorectomy.
* Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy).
* History of bilateral tubal ligation or another surgical sterilization procedure. Approved methods of birth control are as follows: Hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), Tubal Ligation or hysterectomy, Subject/Partner post vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 6 months after completion of RT.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with their ability to safely receive the study interventions are eligible for this trial.
* Ability to understand and the willingness to sign a written informed consent document.

For Arm 1 patients (sinonasal melanoma)

* Patients must have histologically or cytologically confirmed melanoma involving the nasal cavity and/or paranasal sinuses.
* Patients must be evaluated by Head and Neck Surgery to establish surgical status as resectable, borderline resectable or unresectable.
* Patients must have a baseline skull base MRI unless contraindicated by medical or financial toxicity.

For Arm 2 patients (anorectal melanoma)

* Patients must have histologically or cytologically confirmed melanoma involving the anorectal canal.
* Patients must be evaluated by the surgical team to establish primary tumor surgical status as: (1) resectable with sphincter sparing approach, (2) resectable with abdominoperineal resection, or (3) unresectable/requiring surgery greater than abdominoperineal resection.
* Patients must have a baseline rectal MRI unless contraindicated by medical or financial toxicity.

2.2 Exclusion Criteria

* Previous radiation therapy to the planned target area (sinonasal for Arm 1 and anorectal for Arm 2).
* Metastatic disease
* Pregnant women are excluded from this study because RT is a known teratogen.
* Patients who are less than 18 years of age because melanoma is extremely rare in this population and the treatment agent is a known carcinogen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-09-23 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Pathologic Response | through study completion an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Devarati Mitra, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org